CLINICAL TRIAL: NCT03753542
Title: Effect of Nurse-led Education on Parent's Anxiety and Depression on Managing Side Effects of Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nomi Waqas Gul (Other)
Collaborators: Indus Hospital and Health Network (Other)
Responsible Party: Sponsor-Investigator, Nomi Waqas Gul, Principal Investigator, Dow University of Health Sciences
Organization: Dow University of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Enr # 12/2015/912
Record Dates: First submitted 2018-11-16; First posted 2018-11-27 (Actual); Results first posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Chemotherapy Effect
Keywords: chemotherapy, side effects, parents, anxiety, depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Intervention group will received multimedia education, booklet and weekly tele-nursing follow-up about chemotherapy and side effects management
  Interventions: Other: Multimedia education, booklet Providence and tele-nursing follow-up
- Control (No Intervention): The Control group will receive routine care

INTERVENTIONS:
Other: Multimedia education, booklet Providence and tele-nursing follow-up — Multimedia education, booklet and weekly tele-nursing follow-up is about chemotherapy and side effects management
  Arms: Intervention

SUMMARY:
ABSTRACT

Background:

Today, a wide range of pediatric cancers is treated by chemotherapy. More than 21 side effects of chemotherapy have been identified. Among those nausea; vomiting, infection and anemia are most common. The adverse effects are normally managed by the parents at home. Ineffective coping and lack of knowledge about chemotherapy side effect management leads parents stress. Contemporary research evidence that Nurse-led education, booklet providence and follow up about chemotherapy and side effect management, help to decrease parents anxiety and depression.

Objectives:

To measure the effect of nurse-led multimedia education, booklet providence and telephonic follow up about chemotherapy and side effects management on parents anxiety and depression of children receiving chemotherapy for the first time.

Methodology:

A randomized control trial will be conducted in the department of chemotherapy at Indus Children Cancer Hospital Karachi from March 2018 to August 2018 on parents of children below 18 years of age undergoing chemotherapy for the first time. Total 100 parents will be randomly divided into Intervention group (n=50) and Control Group (n=50). The Intervention group will received multimedia education, booklet and weekly tele-nursing follow-up about chemotherapy and side effects management. The Control group will receive routine care. Parent's anxiety and depression will be identified by using DASS-21 and generalized estimating estimation will be used to analyzed the data.

Keywords:

Nurse-led, Multimedia education, Booklet, telephonic follow-up, chemotherapy, side effects, parents, anxiety, depression, children, cancer

DETAILED DESCRIPTION:
INTRODUCTION Background Children Cancer in Pakistan: Millions of people are affected by cancer worldwide. Cancer is one of the major health problems in Pakistan . About 8,000 children below 18 year were diagnosed with cancer annually. Most children diagnosed in advance stage . In Pakistan 31% children had leukemia, 20% had Lymphoma, 08 % had sarcoma, 8 % had bone tumor, 7% had brain tumor, 6 % had retinoblastoma, 5 % had wilms tumor, 4% had germ cell tumor, 4 % had neuroblastoma and the other had 7 % .Cancer affects family emotionally and physically.

Chemotherapy and side effect: Millions of people are also facing difficulties due to chemotherapy worldwide. If the patient will not prepare for chemotherapy treatment properly he/she can face problem in future .Chemotherapy is the common method of treatment. The common side effects of chemotherapy are diarrhea, nausea and vomiting, hair loss, neuropathy, weight loss, dysphagia, oral ulcer, fatigue, dyspnea, constipation, insomnia and cognitive impairment, also affects quality of life, economic conditions, emotions and social wellbeing. Before starting chemotherapy treatment the patient should receive written information about diagnoses, treatment goal, chemotherapy duration, side effects of drugs, the material should design at the level of patient knowledge.

Cancer vs anxiety depression: The anxiety is due to unawareness about chemotherapy side effect. 47% victims of patient have anxiety due to cancer . The power to control disease can be lost due to anxiety .Side effect of chemotherapy management required self-care and it is can be effect due to depression. Anxiety and depression has an association with cancer, chemotherapy related fatigue, lack of education about chemotherapy side effect management and long term exposure of children in hospital . Cancer treatment required nursing intervention to reduce anxiety and depression . Anxiety leads to delay chemotherapy treatment and prognoses.

Evidences of Multimedia education to reduce Anxiety and depression: It is the main responsibility of Oncology nurse to educate patient about the management of side effect of chemotherapy but mostly patient received written material only. The recommended practice to reduce anxiety of patient is to educate about side effect of chemotherapy. The patient should be education both for short term management and long-term management. Education about side effect helps to decrease anxiety. The effect of multimedia education to reduce anxiety is evident in mammography, MRI, ECT, cardiac surgeries, gynecological laparotomy, laparoscopic cystectomy, hemodialysis, teeth removal and peptic ulcer disease. Nursing intervention through education helps to reduce anxiety and stress , after chemotherapy, promote side effect management, decrease complications and increase psychological wellbeing. Many resource centers for patient education on cancer are available on internet about chemotherapy and side effect to increase the psychosocial health. The resources can be utilized as a part of continuous nursing education.

Anxiety and depression in Pakistan: Anxiety and depression is more common in Pakistan due to lack of infrastructure for mental health services.

Aim of the study: The main aim of this study is to find the effect of nurse let chemotherapy education on parent's anxiety as in children case parents are the key role for securing among children cancer. The study will help to examine the effect of psycho-education about chemotherapy and side effect management on parent's anxiety and depression at Indus children cancer Hospital, Karachi Pakistan.

Literature Review

International Findings:

European study found that 20 minutes of video education is more effective with verbal and written education . A randomize control trial was done by Williams and Schreier (2005), on RCT(N=71), the experimental group (n-38) received audiotaped 20 minutes of education on management of fatigue, sleep disturbance and anxiety along with standard care and the control group (n=33) received verbal instruction and written material. The anxiety level was measured at 1 month and 2 months. Larger number of patient (n=16) in control group reported anxiety as compared to experimental group (n=10) significantly (p=0.001). Similar result were found from the study of Malone (2007) that education helps to reduce anxiety. Another study mentioned that familiarity with environment of chemotherapy is necessary as it also impact on anxiety. Almost 50% cases diagnosed with cancer reported the symptoms of anxiety. According to NCCN guideline, the anxiety management related to chemotherapy and side effect management is the primary responsibility of oncology team including oncology nurse . Study from USA mentioned that, the caregiver of children diagnosed with cancer have 44% greater stress as compared to 24% parents of healthy children . Another study mentioned that 98% participant were satisfied with chemotherapy educational experience, 100 % participants mentioned that educational environment is supportive, 81% feel that quality of life can be improved through education . Another study mentioned, 87.6% participant were satisfied with chemotherapy education, 87.5 % agree that it helps to reduce anxiety, 93.3% participant felt that it will be effective if given first time before chemotherapy, 86.6% participant was satisfied for 30 minutes of education timing before chemotherapy treatment. 85.7% participant report that quite room environment is effective for chemotherapy education .In another study mentioned that, 84% patient report that educational class was help to reduce anxiety and 64.7% participant disagree for education in group . A randomize control trail was conducted in Greenville and founded that 23% participant in control group report anxiety after 1 month of treatment as compared to 14% in interventional group significantly . Written information before chemotherapy should be provided to patient, the information should include chemotherapy and side effect, future plan, and follow-up . Many studies had mentioned that that psycho-education is effective to reduce anxiety during chemotherapy management.

Local findings:

A study from Rawalpindi reported that 10-25% participant reported anxiety and depression during chemotherapy and 16% have anxiety and 27% have depression . Another study mentioned that myeloid leukemia is commonly diagnosed in younger age but mostly reported in chronic phase . A study from Lahore mentioned that 56% parents have depression, higher in mothers specially those who are low educated and had poor socio-economical class. A study from Karachi mentioned caregiver stress related to cancer patient s, 17% mild, 34% moderate and 49 % severe stress. It was also conclude that caregiver stress for cancer patient had significant association with caregiver age, relationship with child , female gender and longer duration of care.

Statement of Problem Children cannot look after themselves. Parents are the primary caregiver of children. If they initially feel anxiety and depression, it will be difficult for them to manage chemotherapy and side effects. Education about chemotherapy is neglected due to heavy workload and other responsibilities. More than 50% of individual newly diagnosed with cancer have unknown anxiety related to chemotherapy and their side effect . Those who do not receive chemotherapy education prior to treatment face difficulties in later life . The side effects of chemotherapy like vomiting, nausea, loss of appetite and fatigue were managed through self-care . After an intensive literature review it was found that no study was conducted in Pakistan focusing effect of nurse-led multimedia education and telephonic follow up, on chemotherapy side effects management for parent's anxiety and depression.

Rationale of Study Pediatric cancer is the leading cause of children mortality and morbidity in Pakistan. More than 8,000 children under 18 year of age were diagnosed with cancer in a year. Cancer treatment were managed by the parents specially mother. Evidences showed lack of knowledge about chemotherapy and dissatisfaction of the information about what they have received, leads uncertainty, apprehension and delay continuation with chemotherapy treatment. Many organization developed booklet for patient education about chemotherapy and side effect management. They also have provided online resources. The patient read information at their own efforts. Multimedia education and Tele- nursing follow up was found cost effective method to reduce family anxiety in many countries . Parent's anxiety and depression leads poor management of cancer treatment for their child. Literature evidence that Nurse led psycho-education through multimedia education telephonic follows up is cost effective method to reduce anxiety and depression related to treatment process. According to senior oncologist Pakistan, Parents are anxious not only about Chemo side-effect but also about disease itself. Most parents have same knowledge of side effects of chemotherapy because of their experiences with friend's relatives who have undergo to course treatment. Secondly, side effect is mentioned at first counseling session by primarily oncologist.

Objectives To measure the effect of nurse-led multimedia education, booklet providence and telephonic follow up about chemotherapy and side effects management on parent's anxiety and depression of children receiving chemotherapy for the first time.

Operational Definitions Nurse-Led: Any intervention given by the nurses under professional guidelines. Multimedia education: Education given by using PowerPoint presentation or by using multimedia projector.

Telephonic Follow up: The continuation of educational process by using Tele-communication.

Chemotherapy side effect: The adverse effects of chemotherapy other than therapeutic effect.

Parent's anxiety and depression: Feelings of concern, uneasiness, nervousness and sadness of parents related to child, diagnosed with cancer and undergoing for chemotherapy first time.

ELIGIBILITY:
Inclusion Criteria:

1. Parents along with their Children younger than 18 years of age Note: (Here Child age was taken as Inclusion criteria for Parents, because child age is evident for impact on Parents Psychology, in local study no association of Parents age was evident)
2. Parents along with their children newly diagnosed with cancer in last three weeks
3. Parents along with their children schedule to receive first time chemotherapy in the outpatient department

Exclusion Criteria:

1. Parents along with their children refused to participate
2. Parents along with their children already receiving interventions like multimedia education, booklet providence and telephonic follow up for chemotherapy and side effect management
3. Parents taking medicine for their anxiety and depression. (e.g. Anxiolytics/ Antidepressant)
4. Parents showing uneasiness and discomfort during educational session.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mehwish HUSSAIN, PhD (Statistics), Study Chair — Assistant Professor, DUHS, Karachi; Dr. SHAMVIL ASHRAF, MBBS, DCH, MCPS, FCPS, MRCP, Study Chair — Indus Hospital Karachi; Mr. Hakim Shah, MSN, Study Chair — Associate Professor Institute of Nursing Dow University of Health Sciences Karachi
Locations (1):
- Indus Children Cancer Hospital Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Bhurgri Y, Bhurgri A, Nishter S, Ahmed A, Usman A, Pervez S, Ahmed R, Kayani N, Riaz A, Bhurgri H, Bashir I, Hassan SH. Pakistan--country profile of cancer and cancer control 1995-2004. J Pak Med Assoc. 2006 Mar;56(3):124-30. No abstract available. PMID 16696512
- [Background] Ashraf MS. Pediatric oncology in Pakistan. J Pediatr Hematol Oncol. 2012 Mar;34 Suppl 1:S23-5. doi: 10.1097/MPH.0b013e318249abf9. PMID 22357147
- [Background] CCHK. Children cancer Hospital karachi. 2017 [cited 2017; Available from: http://ccfpakistan.org/.
- [Background] Klein CA. Cancer. The metastasis cascade. Science. 2008 Sep 26;321(5897):1785-7. doi: 10.1126/science.1164853. No abstract available. PMID 18818347
- [Background] Mansoor, S. and S. Jehangir, Anxiety, depression in patient receving chemotherapy for solid tumors. Pak Armed Forces Med. J, 2015. 65(1): p. 89-93.
- [Background] Iqbal A, Siddiqui KS. Depression among parents of children with acute lymphoblastic leukemia. J Ayub Med Coll Abbottabad. 2002 Apr-Jun;14(2):6-9. PMID 12238347
- [Background] Borsellino M, Young MM. Anticipatory coping: taking control of hair loss. Clin J Oncol Nurs. 2011 Jun;15(3):311-5. doi: 10.1188/11.CJON.311-315. PMID 21624866
- [Background] Graca Pereira M, Figueiredo AP, Fincham FD. Anxiety, depression, traumatic stress and quality of life in colorectal cancer after different treatments: A study with Portuguese patients and their partners. Eur J Oncol Nurs. 2012 Jul;16(3):227-32. doi: 10.1016/j.ejon.2011.06.006. Epub 2011 Jul 23. PMID 21783416
- [Background] Pouresmail, Z., S. Sharafi, and M. Razi, The Role of Evidence Based Nursing in Prevention of Gastrointestinal Side Effects of Chemotherapy in Children with Cancer. International Journal of Pediatrics, 2014. 2(2.1): p. 48-48
- [Background] Mohammed, H.A., Impact of proposed nursing rehabilitation program on self management of selected side effects of chemotherapy for elderly patints with gastrointestinal cancer. CU Theses, 2012.
- [Background] Munir F, Burrows J, Yarker J, Kalawsky K, Bains M. Women's perceptions of chemotherapy-induced cognitive side affects on work ability: a focus group study. J Clin Nurs. 2010 May;19(9-10):1362-70. doi: 10.1111/j.1365-2702.2009.03006.x. PMID 20500346
- [Background] Garcia S. The effects of education on anxiety levels in patients receiving chemotherapy for the first time: an integrative review. Clin J Oncol Nurs. 2014 Oct;18(5):516-21. doi: 10.1188/14.CJON.18-05AP. PMID 25164233
- [Background] Hoon LS, Chi Sally CW, Hong-Gu H. Effect of psychosocial interventions on outcomes of patients with colorectal cancer: a review of the literature. Eur J Oncol Nurs. 2013 Dec;17(6):883-91. doi: 10.1016/j.ejon.2013.05.001. Epub 2013 Jun 4. PMID 23759360
- [Background] Lerdkiattikorn, P., et al., Quality of life among stage III colon cancer patients receiving oral and intravenous chemotherapy regimens in Thailand. Mahidol University Journal of Pharmaceutical Sciences, 2012. 39: p. 41-3.
- [Background] Kutlu, R., et al., Kanserli hastalarda depresyon ve yaşam kalitesini etkileyen faktörler. Selçuk Üniv Tıp Derg, 2011. 27(3): p. 149-153
- [Background] Gullatte M. American Society of Clinical Oncology/Oncology Nursing Society chemotherapy safety standards. J Oncol Pract. 2013 Mar;9(2 Suppl):3s-4s. doi: 10.1200/JOP.2012.000862. PMID 24135010
- [Background] Network, N.C.C. Distress management. In NCCN Clinical Practice Guidelines in Oncology. . 2017; Available from: http://www.nccn.org.
- [Background] Leighl N, Gattellari M, Butow P, Brown R, Tattersall MH. Discussing adjuvant cancer therapy. J Clin Oncol. 2001 Mar 15;19(6):1768-78. doi: 10.1200/JCO.2001.19.6.1768. PMID 11251008
- [Background] Williams SA, Schreier AM. The effect of education in managing side effects in women receiving chemotherapy for treatment of breast cancer. Oncol Nurs Forum. 2004 Jan-Feb;31(1):E16-23. doi: 10.1188/04.ONF.E16-E23. PMID 14722602
- [Background] Yasin, Y.M. and A. Al-Hamad, ANXIETY AND DEPRESSION AS KEY DETERMINANTS OF CANCER RELATED FATIGUE AMONG PATIENTS RECEIVING CHEMOTHERAPY. European Scientific Journal, ESJ, 2015. 11(33)
- [Background] Manir KS, Bhadra K, Kumar G, Manna A, Patra NB, Sarkar SK. Fatigue in breast cancer patients on adjuvant treatment: course and prevalence. Indian J Palliat Care. 2012 May;18(2):109-16. doi: 10.4103/0973-1075.100826. PMID 23093826
- [Background] Heidari H, Hasanpour M, Fooladi M. The experiences of parents with infants in Neonatal Intensive Care Unit. Iran J Nurs Midwifery Res. 2013 May;18(3):208-13. PMID 23983756
- [Background] Haugan G, Drageset J. The hospital anxiety and depression scale--dimensionality, reliability and construct validity among cognitively intact nursing home patients. J Affect Disord. 2014 Aug;165:8-15. doi: 10.1016/j.jad.2014.04.042. Epub 2014 Apr 24. PMID 24882171
- [Background] Sarafraz Nasab, M. and M. Mojtabaie, P116: Reminiscence Therapy Efficacy in Reducing Symptoms of Anxiety in Elderly Nursing Home Residents in Tehran. The Neuroscience Journal of Shefaye Khatam, 2014. 2(3): p. 140-140.
- [Background] Zakerimoghadam, M., S. Ghiasvandian, and P. Salahshoor, The effect of supportive nursing program on depression, anxiety and stress of family members of patients during coronary artery bypass graft (CABG) surgery. Iranian Journal of Cardiovascular Nursing, 2014. 3(1): p. 50-58

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The parents along with children were recruited in the study from September 2018 to November 2018 and follow up were continued from October 2018 to December 2018. After the completion of follow up to 5th December 2018 the trail was ended due to the completion of target sample sized (N=100) of parents and follow up schedule.The age of children were taken as associated factor for parent as study evident that children age has impact on parents anxiety. Parent age was not taken due to guardian issue.
Pre-assignment Details: Total 100 parents were randomly divided into Intervention group (n=50) and Control Group (n=50). After excluding lost to follow up, the data was analyzed from 77 sample of parents (41 in intervention group and 36 in control group). The intervention group received multimedia education, booklet and weekly tele-nursing follow-up about chemotherapy and side effects management. The control group received routine care.
Groups:
- Intervention: The Intervention group received multimedia education, booklet and weekly tele-nursing follow-up about chemotherapy and side effects management
- Control: The Control group receive routine care
Period: Overall Study
Arm/Group | Intervention | Control
Started | 50 (Actual Calculated Sample size was 30 Sample, 100 was taken to restore lost to follow up) | 50 (Actual Calculated Sample size was 30 Sample, 100 was taken to restore lost to follow up)
Completed | 41 (In spite of having lost to follow up the power of study was not lost) | 36 (In spite of having lost to follow up the power of study was not lost)
Not Completed | 9 | 14
Not completed — Lost to Follow-up | 9 | 14

BASELINE CHARACTERISTICS:
Population: After excluding lost to follow up total data analyse in intervention group was 41 and control group was 36
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 41 | 36 | 77
Age, Customized [Count of Participants; unit: Participants] — Note: In this study age of children were taken as associated factor for parents anxiety, depression and stress because local studies evident that age of children were associated with parent psychology. The age of parent were not assess due to guardian issues. It is recommended, other student should also take the age of parents. As the age of parents was not taken hence it may be considered as limitations in this study.
  Participants
    1. Child Age:: 2-4years | 13 | 11 | 24
    1. Child Age:: 5-7years | 10 | 8 | 18
    1. Child Age:: 8-12 years | 12 | 12 | 24
    1. Child Age:: 13-18 years | 6 | 5 | 11
Sex/Gender, Customized [Count of Participants; unit: Participants] — In this study Gender of the children were assessed instead gender of the parents, because gender discrimination e.g Male child Vs Female child is common at local level. Gender of children has psychological effect on parents. e.g. Male children support family while female not. This type of thinking is common in Poor socioeconomic situation. Gender of parents were not taken due to guardian issues. Other studies are recommended to take gender of the parent as associative factors.
  Participants
    2. Child Gender:: Male | 24 | 26 | 50
    2. Child Gender:: Female | 17 | 10 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
3. Primary Care Giver: [Count of Participants; unit: Participants]
  Mother/Father | 38 | 30 | 68
  Others | 3 | 6 | 9
4. Residency/Locality: [Count of Participants; unit: Participants]
  Local | 17 | 11 | 28
  Non- Local | 24 | 25 | 49
5. Occupation [Count of Participants; unit: Participants]
  Labor | 24 | 18 | 42
  Shopkeeper | 8 | 9 | 17
  Other | 9 | 9 | 18
6. Level of education [Count of Participants; unit: Participants]
  Uneducated | 11 | 11 | 22
  School Education | 17 | 16 | 33
  Higher Education | 13 | 9 | 22
7. Employment status [Count of Participants; unit: Participants]
  Daily Wages | 28 | 21 | 49
  Monthly Salary | 13 | 15 | 28
8. Income per month (Rupees) [Count of Participants; unit: Participants]
  less than 10,000 | 12 | 17 | 29
  More than 10,000 | 29 | 19 | 48
9 Child Diagnoses [Count of Participants; unit: Participants]
  Leukemia | 28 | 23 | 51
  Other | 13 | 13 | 26
10. Family History of cancer [Count of Participants; unit: Participants]
  No | 34 | 33 | 67
  Yes | 7 | 3 | 10
11. Pain felt by the child [Count of Participants; unit: Participants]
  No | 23 | 26 | 49
  yes | 18 | 10 | 28
12. Do parent have smoking habits? [Count of Participants; unit: Participants]
  No | 21 | 23 | 44
  Yes | 20 | 13 | 33
Depression [Mean (Standard Deviation); unit: units on a scale] | 15.41 (5.97) | 16.28 (7.32) | 15.82 (6.6)
Anxiety [Mean (Standard Deviation); unit: units on a scale] | 11.9 (6.51) | 10.72 (7) | 11.35 (6.72)
Stress [Mean (Standard Deviation); unit: units on a scale] | 16.63 (5.96) | 16.67 (6.45) | 16.65 (6.15)

OUTCOME MEASURES:

1. Primary Outcome: Depression, Anxiety and Stress Scale - 21 (DASS-21)
Description: DASS-21 is comprised of questionnaires for three separate scales measuring Depression, Anxiety and Stress. The depression scale is scored by summing the responses of each question, multiplying by 2 and then scoring on a scale ranging from a minimum of 0 to a maximum of 28+, with higher scores indicating greater severity. The anxiety scale is scored by summing the responses of each question, multiplying by 2 and then scoring on a scale ranging from a minimum of 0 to a maximum of 20+, with higher scores indicating greater severity. The stress scale is scored by summing the responses of each question, multiplying by 2 and then scoring on a scale ranging from a minimum of 0 to a maximum of 37+, with higher scores indicating greater severity
Time Frame: up to 4 weeks
Population: Total 100 parents were enrolled and randomly allocated to (i)intervention group and (ii)Control group with equal number of allocations in each group respectively. The data were analyzed after excluding lost to follow up variables.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: The Control group will receive routine follow up.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 41 | 36
score on a scale
  Post-Depression (After 1 week) | 6.44 (3.94) | 9.72 (5.82)
  Two- Week Post Depression (After 2 week) | 2.63 (2.98) | 6.11 (4.94)
  Post-Anxiety (After 1 week) | 4.2 (3.43) | 6.61 (5.23)
  Two- Week Post Anxiety (After 2 week) | 1.75 (2.33) | 4.27 (3.61)
  Post-Stress (After 1 week) | 7.02 (4.59) | 11 (6.3)
  Two- Week Post Stress (After 2 week) | 2.88 (3.1) | 6.83 (5.22)

ADVERSE EVENTS:
Time Frame: 2 months
Description: The intervention were limited to Parents education only. . The education was given under international guideline of NIH. Hence, Adverse Events were not monitored/assessed/ nor reported by participant.
Groups:
- Intervention; Control: No Adverse event reported
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
As the study was conducted in single setting, hence the result may not be generalized. Further studies are recommended to measure its general effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT03753542/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT03753542/ICF_001.pdf